CLINICAL TRIAL: NCT02891395
Title: Efficacy and Safety of Nilotinib in Patients With a Chronic Disease of the Graft Against the Host (Graft Versus Host, GVH) Did Not Respond to Imatinib Mesylate.
Brief Title: Efficacy and Safety of Nilotinib in Patients With a Chronic Disease of the Graft Against the Host
Acronym: DoubleITK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009_18; 2012-000770-36 (EudraCT Number)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2019-07

CONDITIONS: Graft Versus Host Disease
Keywords: allogeneic stem cell transplantation; imatinib Mesylate; Nilotinib
MeSH Terms: conditions — Graft vs Host Disease | interventions — Imatinib Mesylate; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open-label (Experimental): Induction phase: Imatinib mesylate - starting with 100 mg/day with increase of 100 mg/day each other week up to maximum tolerable dose or 400 mg/day whichever occurred first. For the responders and in absence of toxicity, the treatment will be maintained up to one year.
  Salvage phase:
  Nilotinib - starting with 200 mg/day with increase of 200 mg/day each other week up to maximum tolerable dose or 800 mg/day whichever occurred first. In absence of toxicity, the treatment will be maintained up to one year.
  Interventions: Drug: Imatinib Mesylate and Nilotinib

INTERVENTIONS:
Drug: Imatinib Mesylate and Nilotinib — For patients under Imatinib Mesylate: the total length of follow up period for those patients will be for 52 weeks following IM treatment, with a follow up at weeks IM4, IM8, IM12, IM26, IM38 and IM52.
  For patients requiring a salvage phase: after the switch for nilotinib, the total length of follow up period for this phase will be for 52 weeks following nilotinib treatment, with a follow up at weeks nilo4, nilo8, nilo12, nilo26, nilo38 and nilo52.

SUMMARY:
Open label non-randomized multicenter phase 2 trial with direct individual benefice

DETAILED DESCRIPTION:
Induction phase: Imatinib mesylate - starting with 100 mg/day with increase of 100 mg/day each other week up to maximum tolerable dose or 400 mg/day whichever occurred first. For the responders and in absence of toxicity, the treatment will be maintained up to one year. Patients, who discontinue imatinib mesylate at 3 months for lack of response (no response = stable disease), those who experience progression at any time, those who relapse after an initial response at any time or those who discontinue for toxicity at any time, will go to the salvage phase.

Salvage phase:

Nilotinib - starting with 200 mg/day with increase of 200 mg/day each other week up to maximum tolerable dose or 800 mg/day whichever occurred first. In absence of toxicity, the treatment will be maintained up to one year.

ELIGIBILITY:
Inclusion Criteria:

Induction phase (IM):

* Patients aged ≥18 years to 75 years
* Patients who underwent allo-SCT for a hematological disorder
* Body weight ≥ 40 Kg.
* Confirmed diagnosis of cGVHD resistant to at least one systemic immunosuppressive therapy. The diagnosis of cGHVD should be based on the NIH Working Group Consensus (www.asbmt.org/gvhd/index.htm). Grading of cGVHD will be based on clinical manifestations including:

  1. ocular, oral and mucosal symptoms;
  2. performance status;
  3. evaluation of pulmonary functions;
  4. cutaneous evaluation;
  5. evaluation of musculo-skeletal manifestations;
  6. evaluation of liver involvement;
* Any source of hematopoietic stem cell is allowed
* Both myeloablative and nonmyeloablative conditioning regimens are authorized.
* Absence of contra-indications to the use of IM or Nilotinib
* Patient having French health care coverage
* Female patients of childbearing potential must have before initiation of study drug and agree to have efficient contraceptive precautions throughout the trial and for 3 months after the end of the trial.
* Signed informed consent.

Salvage phase (Nilotinib) :

Patients enrolled in the first phase and who failed to IM:

* Patients, who discontinue imatinib mesylate at 3 months for lack of response (no response = stable disease),
* those who experience progression at any time,
* those who relapse after an initial response at any time
* or those who discontinue for toxicity at any time.

Exclusion Criteria:

* Patient developing acute GVHD (whether early or "late onset" form)
* First episode of cGVHD
* Patient who received IM or Nilotinib treatment or any other TKI after transplant 3 months before the inclusion on the study
* Patient treated by TKI for a GVHD
* Contra-indication to IM or Nilotinib
* Neutropenia < 0.5 G/L
* Uncontrolled systemic infection which can be associated, according to the investigator, to an enhanced risk of patient's death during the first month of treatment
* Severe neurological or psychiatric disorders
* Pregnancy or lactation
* Known uncontrolled arrhythmias or symptomatic heart disease or left ventricular ejection fraction < 40% (cardiac tests as clinically indicated)
* Recurrence of cancer for which the transplant was done except for presence of minimal residual disease by PCR
* Patients with secondary malignancy ≤ 2 years prior study-entry except:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Prostate cancer (Tumor, Node, Metastasis [TNM] stage T1a or T1b)
* Patients in emergency situation
* Patients kept in detention
* Patients unable or unwilling to comply with the protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-12-24 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Response rate at 3 months (complete and partial remission) after salvage treatment with Nilotinib in patients with chronic GVHD who failed Imatinib Mesylate (IM) | Between Baseline and minimum 12 weeks of treatment
  Response rate at 3 months (complete and partial remission) after salvage treatment with Nilotinib in patients with chronic GVHD who failed Imatinib Mesylate (IM)

SECONDARY OUTCOMES:
Best response to IM within 12 months and the duration of this response | From 12 to 52 weeks of Imatinib Mesylate treatment
Best response rate to Nilotinib within 12 months and the duration of this response | From 12 to 52 weeks of Nilotinib treatment
use of systemic secondary treatment due to intolerance to IM | From baseline to 12 weeks of IM treatment
  measure intolerance by IM failure
use of systemic secondary treatment due to intolerance to Nilotinib | From baseline to 12 weeks of Nilotinib treatment
  measure intolerance by Nilotinib failure

CONTACTS AND LOCATIONS:
Overall Officials: YAKOUB-AGHA Ibrahim, MD, Principal Investigator — University Hospital, Lille
Locations (22):
- CHU Sart Tilman, Liège, Belgium
- France (21):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - Hopital Morvan, Brest
  - CHU Clémenceau, Caen
  - HIA de Percy, Clamart
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Diseases of Blood Service HURIEZ hospital CHRU de LILLE, Lille
  - Centre hospitalier et régional de Lille, Lille
  - CHU de Lyon, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Saint Eloi, Montpellier
  - CHU Hotel Dieu, Nantes
  - CHU de Nice, Nice
  - Hopital NECKER, Paris
  - Hôpital pitié Salpetrière, Paris
  - Centre Henri Becquerel, Rouen
  - CHU de STRASBOURG, Strasbourg
  - CHU Purpan, Toulouse

REFERENCES:
- [Result] Srour M, Alsuliman T, Labreuche J, Bulabois CE, Chevallier P, Daguindau E, Forcade E, Francois S, Guillerm G, Coiteux V, Turlure P, Beguin Y, Yakoub-Agha I, Magro L. Nilotinib efficacy and safety as salvage treatment following imatinib intolerance and/or inefficacy in steroid refractory chronic graft-versus-host-disease (SR-cGVHD): a prospective, multicenter, phase II study on behalf of the Francophone Society of Bone Marrow Transplantation and Cellular Therapy (SFGM-TC). Bone Marrow Transplant. 2023 Apr;58(4):401-406. doi: 10.1038/s41409-022-01898-x. Epub 2023 Jan 9. PMID 36624161